CLINICAL TRIAL: NCT06169670
Title: Prospective Evaluation of Autologous Fat Grafting to the Face With the Use of Viality™ in Processing of Lipoaspirate
Brief Title: Autologous Fat Grafting to the Face With Use of the Viality™ System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tiger Biosciences, LLC. (Industry)
Collaborators: Faces+ (Other)
Responsible Party: Principal Investigator, Steven Cohen, Plastic Surgeon, Tiger Biosciences, LLC.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VIAL-001
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Adipose Tissue
Keywords: fat transfer; Viality; Injectable Tissue Replacement and Regeneration; midfacial

STUDY DESIGN:
Intervention Model Description: This is a single-center, prospective study enrolling patients undergoing an aesthetic fat grafting procedure to the face. A total of 20 patients will be enrolled in the study, all patients will receive lipoaspirate processed with Viality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Patients Receiving Lipoaspirate with Viality (Experimental): Patient will be undergoing fat transfers to the face with lipoaspirate processed using the Viality wash system.
  Interventions: Device: Viality

INTERVENTIONS:
Device: Viality — Viality is a lipoaspirate wash system designed to be used in the operating room in conjunction with, and attached to, a user-provided liposuction cannula, a vacuum source, and a waste canister.
  Viality is to be used to filter and wash aspirated, harvested autologous adipose tissue for aesthetic body contouring. The system should be used with a legally marketed vacuum or aspirator apparatus as a source of suction. If harvested fat is to be re-implanted, the harvested fat is to be used without any additional manipulation. Viality is not intended to process autologous adipose tissue other than for aesthetic body contouring uses.

SUMMARY:
The purpose of this research is to collect data on the short and long-term effects of facial fat grafting by injectable tissue replacement and regeneration in the midfacial zone, with the use of the VialityTM system. The Viality system is a US Food and Drug Administration (FDA) cleared device.

DETAILED DESCRIPTION:
Autologous fat transfer (AFT) is a minimally invasive medical procedure that includes aspirating adipose tissue from one part of the body and washing, filtering, and reinjecting the processed fat tissue into a different part of the body with the primary purpose of adding volume.

A 2013 survey of the American Society of Plastic Surgeons indicated that 80% of the responding physicians use AFT.

Several published studies conclude that using a filter mesh to concentrate the fat by removing surgical tumescent fluid and blood improves fat graft retention (Salinas et al., Girard et al., Ansorge et.al.). Furthermore, washing and filtration of the autologous adipose tissue produces a fat graft with higher tissue viability (Zhu et al., Girard et al., Barbour et al.)

Viality is a lipoaspirate wash system designed to be used in the operating room in conjunction with, and attached to, a user-provided liposuction cannula, a vacuum source, and a waste canister.

Viality is to be used to filter and wash aspirated, harvested autologous adipose tissue for aesthetic body contouring. The system should be used with a legally marketed vacuum or aspirator apparatus as a source of suction. If harvested fat is to be re-implanted, the harvested fat is to be used without any additional manipulation. Viality is not intended to process autologous adipose tissue other than for aesthetic body contouring uses.

ELIGIBILITY:
Inclusion Criteria:

* Female patients > 18 years and < 65 years of age.
* Patients undergoing an aesthetic fat grafting procedure to the face.
* Patients must be able to provide written informed consent, understand and be willing to comply with study-related procedures and follow-up visits.
* Patients must be non-smokers.
* Patients with available/adequate harvest sites for fat grafting.
* Anticipated harvested fat volume between 60 and 100 cc.
* Anticipated fat injection volume 40-55 cc.
* Patients must agree to maintain their weight (i.e. within 5%) by not making any major changes in diet or lifestyle during the study.

Exclusion Criteria:

* Skin rash in the treatment area.
* Patients who smoke or use nicotine products.
* Patients with bleeding disorders or currently taking anticoagulants.
* Patients with history of trauma or surgery to the treatment area.
* Active, chronic, or recurrent infection.
* Compromised immune system.
* Hypersensitivity to analgesic agents.
* Co-morbid condition that could limit ability to participate in the study or to comply with follow-up requirements.
* Untreated drug and/or alcohol abuse.
* Pregnant or breastfeeding.
* Any issue that, at the discretion of the investigator, would contra-indicate the patient's participation.
* Patients who do not wish to have the study area photographed.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female patients who are not and do not plan to be pregnant or breastfeeding during the duration of the study.
Enrollment: 20 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2025-01-13 (Estimated); Study Completion 2025-03-13 (Estimated)

PRIMARY OUTCOMES:
Facial Fat Volume Retention | 12 months
  Facial fat volume retention after facial fat transfer using Viality system will be monitored over the course of year and retrospectively compared to facial fat volume retention after facial fat transfers using traditional fat processing.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Saul, Study Director — Coordinator
Locations (1):
- Faces Plus, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: Yes
The Sponsor will also monitor the site at various intervals. Case Report Forms and Investigator Binders will be reviewed for current data.
Time Frame: The Sponsor will collect data once patients have been followed for 3 months, 6 months, and at the end of the 12 month follow-up period.
Access Criteria: Investigators with permission from the Primary Investigator or the Sponsor will be granted access to patient files stored on a secured server.